CLINICAL TRIAL: NCT01912963
Title: A Phase II Study of Eribulin Mesylate in Combination With Trastuzumab and Pertuzumab in Women With Metastatic, Unresectable Locally Advanced, or Locally Recurrent Human Epidermal Growth Factor Receptor 2-Positive Breast Cancer
Brief Title: Phase II Study of Eribulin Mesylate, Trastuzumab, and Pertuzumab in Women With Metastatic, Unresectable Locally Advanced, or Locally Recurrent HER2-Positive Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study terminated early due to weak accrual.
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Eisai Inc. (Industry); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Rachel Freedman, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-163
Record Dates: First submitted 2013-07-24; First posted 2013-07-31 (Estimated); Results first posted 2018-12-05 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-11

CONDITIONS: HER2-positive Breast Cancer; Metastatic Breast Cancer
Keywords: HER-2 Positive Breast Cancer; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pertuzumab; Trastuzumab; eribulin

STUDY DESIGN:
Intervention Model Description: Of note, this is not a parallel assignment rather one Phase I arm and two Phase II arms all independently evaluated.
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Phase I: Dose Level 1 (D1) (Experimental): Pertuzumab: 840 mg/cycle 1 then 420 mg/cycle IV on day 1
  Trastuzumab: 8 mg/kg/cycle 1 then 6 mg/kg cycle IV on day 1
  Eribulin: 1.4 mg/m2/cycle IV on days 1 and 8 (D1)
  Cycle duration=21 days
  The Phase I run-in potentially evaluates 2 dose levels of eribulin in combination with pertuzumab and trastuzumab. Participants first receive antibody administration then eribulin. In the treatment phase, participants receive up to 6 cycles of combination therapy unless disease progression (PD) or withdrawal for other reasons (w/d). Participants who complete 6 cycles have the option to continue with antibody therapy only until PD or w/d in the extension phase.
  Interventions: Drug: Pertuzumab; Drug: Trastuzumab; Drug: eribulin
- Phase II Cohort A: Without Prior Pertuzumab Exposure (Experimental): Pertuzumab: 840 mg/cycle 1 then 420 mg/cycle IV on day 1
  Trastuzumab: 8 mg/kg/cycle 1 then 6 mg/kg cycle IV on day 1
  Eribulin: 1.4 mg/m2/cycle IV on days 1 and 8 (recommended phase II dose)
  Cycle duration=21 days
  In the Phase II study, participants enrolled into two possible cohorts based on prior pertuzumab exposure. Participants first receive antibody administration then eribulin. In the treatment phase, participants receive up to 6 cycles of combination therapy unless disease progression (PD) or withdrawal for other reasons (w/d). Participants who complete 6 cycles have the option to continue with antibody therapy only until PD or w/d in the extension phase.
  Interventions: Drug: Pertuzumab; Drug: Trastuzumab; Drug: eribulin
- Phase II Cohort B: With Prior Pertuzumab Exposure (Experimental): Pertuzumab: 840 mg/cycle 1 then 420 mg/cycle IV on day 1
  Trastuzumab: 8 mg/kg/cycle 1 then 6 mg/kg cycle IV on day 1
  Eribulin: 1.4 mg/m2/cycle IV on days 1 and 8 (recommended phase II dose)
  Cycle duration=21 days
  In the Phase II study, participants enrolled into two possible cohorts based on prior pertuzumab exposure. Participants first receive antibody administration then eribulin. In the treatment phase, participants receive up to 6 cycles of combination therapy unless disease progression (PD) or withdrawal for other reasons (w/d). Participants who complete 6 cycles have the option to continue with antibody therapy only until PD or w/d in the extension phase.
  Interventions: Drug: Pertuzumab; Drug: Trastuzumab; Drug: eribulin

INTERVENTIONS:
Drug: Pertuzumab
  Other Names: Perjeta
Drug: Trastuzumab
  Other Names: Herceptin
Drug: eribulin
  Other Names: eribulin mesylate; Halaven

SUMMARY:
In this study, the investigators are testing the effectiveness of the combination of eribulin, pertuzumab and trastuzumab to learn whether this combination of drugs works in treating advanced HER2-positive breast cancer that had received at least one prior treatment previously. At this point, the standard treatment for HER2-positive cancer that has progressed (grown) after a first treatment is chemotherapy combined with therapies that target the HER2 protein (e.g., trastuzumab or lapatinib).

DETAILED DESCRIPTION:
All of the medications that are being tested in this study are approved by the Food and Drug administration (FDA) for the treatment of metastatic breast cancer. However, the combination of these three medications in participants has not yet been tested. Eribulin is a chemotherapy agent that is approved for the treatment of metastatic breast cancer for women who have previously received at least two prior chemotherapeutic regimens for the treatment of their metastatic disease. Pertuzumab and trastuzumab are also both approved for the treatment of advanced HER2-positive breast cancer. Both agents help treat breast cancer by binding HER2 receptor. However, pertuzumab and trastuzumab bind to different parts of the HER2 receptor. Another scientific goal of this research study is to perform gene sequencing (gene tests) on your cancer cells (obtained from biopsies or surgery) and normal tissues (usually blood). The results of the gene tests will be used to try to develop better ways to treat and prevent cancers.

After the Phase I run-in, two cohorts based on prior exposure to pertuzumab were evaluated. The target accrual for Cohort A, without prior pertuzumab, is 56 participants. Using a two-stage design (n=34 stage 1, n=22 stage 2), there is 90% power assuming 10% Type I error to determine whether objective response (OR) rate is consistent with the alternative rate of 40% versus the null rate of 24%. There is 57% probability of stopping the trial at stage one if the true OR rate is 24%. Cohort B, with prior pertuzumab, is evaluated using a single stage design. There is 91% power to detect an improvement in OR from 10% to 30% with accrual of 25 participants.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet the following criteria on screening examination to be eligible to participate in the study:

- Participants must have invasive primary tumor or metastatic tissue confirmation of human epidermal growth factor receptor 2 (HER2)-positive status, defined as presence of one or more of the following criteria: Over-expression by immunohistochemistry (IHC) with score of 3+ AND/OR HER2 gene amplification (> 6 HER2 gene copies per nucleus or a FISH ratio [HER2 gene copies to chromosome 17 signals] of ≥ 2.0) Note: Participants with a negative or equivocal overall result (FISH ratio of <2.0 or ≤ 6.0 HER2 gene copies per nucleus) and IHC staining scores of 0, 1+, 2+ are not eligible for enrollment.

* Participants must have metastatic, unresectable locally advanced, or locally recurrent HER2-positive breast cancer. For the phase II portion of the study, it is required that participants have measurable disease, as defined by RECIST 1.1, which can be accurately evaluated on computerized tomography (CT) or magnetic resonance (MRI). Measurable disease is defined as: at least one lesion of >10 mm in the longest diameter for a non-lymph node or >15 mm in the short-axis diameter for a lymph node which is serially measurable according to RECIST 1.1.criteria.1
* Participants must have received at least 1 line of chemotherapy for advanced or metastatic breast cancer and/or relapse/progressed while on or within 6 months of completion of neoadjuvant or adjuvant trastuzumab. Prior pertuzumab is allowed in the phase II portion of the trial.
* Participants must have had prior trastuzumab therapy (either in the adjuvant or metastatic setting).
* Participants must be at least 2 weeks out from prior endocrine therapy, chemotherapy,radiotherapy, or other cancer-directed therapy (including novel agents), with adequate recovery of toxicity to baseline, or grade ≤1, with the exception of alopecia and hot flashes. Participants may have initiated bisphosphonate/denosumab therapy prior to start of protocol therapy. Biphosphonate/denosumab therapy may continue during protocol treatment. Such participants will have bone lesions considered evaluable for progression. Washout for trastuzumab is not necessary.
* Women and men, age 18 years at the time of informed consent.
* Participants must have an Eastern Cooperative Oncology Group (ECOG) performance status 0-1 or a Karnofsky Performance Scale (KP) 70%.
* Participants must have normal organ and marrow function as defined below:
* Absolute neutrophil count > 1,500/mcL
* Platelets > 75,000/mcL
* Hemoglobin >9g/dl
* Total bilirubin ≤2.0 X institutional upper limit of normal
* Aspartate Aminotransferase (AST, SGOT)/ALT(Alanine Aminotransferase, SGPT) ≤ 3 X institutional ULN without liver metastases, or ≤ 5 times institutional upper limit normal (ULN) with liver metastases (if liver metastases felt to be cause of Liver function tests (LFT) abnormalities)
* Alkaline phosphatase (ALP) ≤3 x institutional upper limit of normal If total ALP is >3x institutional upper limit normal (in the absence of liver metastasis) or >5x institutional upper limit of normal (in subjects with liver metastasis) AND the subject is known to have bone metastases, then liver ALP isoenzyme should be used to assess liver function rather than total ALP.
* Creatinine 2.0 mg/dL or creatinine clearance ≥50 mL/min.
* left ventricular ejection fraction (LVEF) ≥50%, as determined by radionucleoventilugrams (RVG) (multi-gated acquisition-MUGA) or Echocardiogram (ECHO) within 60 days prior to initiation of protocol therapy.
* Adequate IV access
* The effects of eribulin mesylate, trastuzumab, and pertuzumab on the developing human fetus are unknown. Pre-clinical data was suggestive of a teratogenic effect of eribulin mesylate. Pertuzumab caused oligohydramnios, delayed renal development and embryo-fetal deaths in pregnant cynomolgus monkeys. In the post-marketing setting, cases of oligohydramnios, some associated with fatal pulmonary hypoplasia of the fetus have been reported in pregnant women receiving trastuzumab. For these reasons women of child bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and willingness to sign a written informed consent document (approved by Institutional review board or independent ethics committee) obtained prior to any study procedure, with the understanding that the subject may withdraw at any time without prejudice.
* Laboratory tests required for eligibility must be completed within 14 days prior study entry. Baseline tumor measurements must be documented from tests within 28 days of study entry. Other non-laboratory tests must be performed within 28 days of study entry.
* For the Phase 2 portion of the study; patients must have tissue that is amenable to biopsy and must be willing to undergo research biopsy.

Exclusion Criteria: - Participants who exhibit any of the following conditions at screening will not be eligible for admission into the study:

* Participants receiving any other study agents.
* Participants receiving any other cancer directed concurrent therapy; such as concurrent chemotherapy, radiotherapy, or hormonal therapy. Concurrent treatment with biphosphonates/denosumab is allowed but should be started before starting treatment on study.
* Active brain metastases: Participants with previously diagnosed brain metastases are eligible if they have completed treatment at least one month prior to enrollment, are neurologically stable, and have recovery from effects of radiotherapy or surgery.
* History of allergic reaction attributed to compounds of similar chemical or biologic composition to eribulin mesylate, trastuzumab or pertuzumab, which cannot be managed by premedication.
* Participants who previously received eribulin mesylate are not eligible for enrollment on the phase II portion.
* Prior chemotherapy, targeted therapy, hormonal therapy, or radiation therapy (including any investigational agents) within 2 weeks prior entering the study or those who have not recovered adequately from adverse events (AEs) due to agents administered more than 4 weeks earlier (excluding alopecia and hot flashes). A washout period is not necessary for trastuzumab (or pertuzumab for run-in patients when applicable).
* A baseline corrected QT interval of > 470 ms.
* Pre-existing neuropathy ≥ grade 2 (NCI Common Toxicity Criteria for Adverse Events (CTCAE) Version 4.0)
* Uncontrolled intercurrent illness including, not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements or other significant diseases or disorders that, in the investigator's opinion, would exclude the subject from participating in the study
* Symptomatic intrinsic lung disease or extensive tumor involvement of the lungs, resulting in grade 2 or higher dyspnea at rest.
* Currently pregnant or breast-feeding. All females must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of β-Human Chorionic Gonadotropin (β-Hcg) at the Baseline visit [within 7 days of the first dose of study treatment]). Females of childbearing potential must agree to use a medically acceptable method of contraception (e.g., abstinence, an intrauterine device, a double-barrier method such as condom + spermicidal or condom + diaphragm with spermicidal, a contraceptive implant, an oral contraceptive or have a vasectomized partner with confirmed azoospermia) throughout the entire study period and for 30 days after discontinuation of study treatment. The only subjects who will be exempt from this requirement are postmenopausal women (defined as women who have been amenorrheic for at least 12 consecutive months, in the appropriate age group, without other known or suspected primary cause) or subjects who have been sterilized surgically or who are otherwise proven sterile (i.e., bilateral tubal ligation with surgery at least 1 month before start of study treatment, hysterectomy, or bilateral oophorectomy with surgery at least 1 month before start of study treatment). Current, ongoing protocols containing pertuzumab have included continuous pregnancy monitoring during the trial and for six months after the last dose of study drug is administered. Because of the long half-life of pertuzumab, women should be warned not to become pregnant for at least six months after completion of treatment.
* Individuals with a history of different malignancy are ineligible except for the following circumstances. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: cervical cancer in situ, and non-melanoma cancer of the skin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Freedman, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Balch SM, Vaz-Luis I, Li T, Tayob N, Jain E, Helvie K, Buendia-Buendia JE, Shannon E, Isakoff SJ, Tung NM, Krop IE, Lin NU, Wagle N, Freedman RA. A phase II study of efficacy, toxicity, and the potential impact of genomic alterations on response to eribulin mesylate in combination with trastuzumab and pertuzumab in women with human epidermal growth factor receptor 2 (HER2)+ metastatic breast cancer. Breast Cancer Res Treat. 2021 Sep;189(2):411-423. doi: 10.1007/s10549-021-06329-x. Epub 2021 Jul 24. PMID 34302589
- See also: American Society Clinical Oncology (ASCO) 2017 abstract — http://ascopubs.org/doi/abs/10.1200/JCO.2017.35.15_suppl.1034

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled from September 2013 through May 2016.
Groups:
- Phase II Cohort B: With Prior Pertuzumab Exposure: Pertuzumab: 840 mg/cycle 1 then 420 mg/cycle IV on day 1
  Trastuzumab: 8 mg/kg/cycle 1 then 6 mg/kg cycle IV on day 1
  Eribulin: 1.4 mg/m2/cycle IV on days 1 and 8 (recommended phase II dose)
  Cycle duration=21 days
  In the Phase II study, participants enrolled into two possible cohorts based on prior pertuzumab exposure. Participants first receive antibody administration then eribulin. In the treatment phase, participants receive up to 6 cycles of combination therapy unless disease progression (PD) or withdrawal for other reasons (w/d). Participants who complete 6 cycles have the option to continue with antibody therapy only until PD or w/d in the extension phase.
  Pertuzumab
  Trastuzumab
  eribulin
Period: Overall Study
Arm/Group | Phase I: Dose Level 1 (D1) | Phase II Cohort A: Without Prior Pertuzumab Exposure | Phase II Cohort B: With Prior Pertuzumab Exposure
Started | 6 | 19 | 7
Completed (Since treatment was not of fixed duration, all participants were considered 'Not Completed'.) | 0 | 0 | 0
Not Completed | 6 | 19 | 7
Not completed — Disease Progression (RECIST1.1) | 6 | 9 | 5
Not completed — Disease Progression (not RECIST1.1) | 0 | 7 | 1
Not completed — Adverse Event | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Sought treatment locally | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The analysis dataset is comprised all enrolled patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I: Dose Level 1 (D1) | Phase II Cohort A: Without Prior Pertuzumab Exposure | Phase II Cohort B: With Prior Pertuzumab Exposure | Total
Number analyzed (Participants) | 6 | 19 | 7 | 32
Age, Continuous [Median (Full Range); unit: years] | 55 [38 to 66] | 53 [33 to 73] | 47 [40 to 70] | 53 [33 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 19 | 7 | 31
  Male | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 2
  White | 6 | 14 | 7 | 27
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 0 | 3
Region of Enrollment [Number; unit: count of participants]
  United States | 6 | 19 | 7 | 32
Time from Primary Diagnosis to metastatic diagnosis [Number; unit: count of participants]
  < 2 years | 1 | 5 | 4 | 10
  > 2 years | 2 | 8 | 2 | 12
  Metastatic diagnosis at primary diagnosis | 3 | 6 | 1 | 10
ECOG PS [Number; unit: count of participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) ECOG PS 0: Fully active, able to carry on all pre-disease performance without restriction ECOG PS 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature ECOG PS 2: Ambulatory and capable of all self-care but unable to carry out any work activities; Up and about more than 50% of waking hours
  count of participants
    ECOG PS 0 | 5 | 14 | 4 | 23
    ECOG PS 1 | 1 | 4 | 3 | 8
    Unknown | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Eribulin the Recommended Phase II Dose (RP2D) [Phase I]
Description: The RP2D of eribulin in combination with pertuzumab and trastuzumab is determined by the number of patients who experience a dose limiting toxicity (DLT). See subsequent primary outcome measure for the DLT definition. The RP2D is defined as the highest dose at which fewer than one-third of six patients experience a DLT. In this Phase I run-in, only 2 dose levels were under evaluation: a starting dose (D1) and a de-escalation dose (D-1) if 2 or more DLTs are observed in Dose Level 1 (DL1).
Time Frame: The observation period for the RP2D was the 1st cycle of treatment.
Population: The analysis dataset is comprised all enrolled Phase I participants.
Measure: Number; unit: mg/m^2
Groups:
- Phase I: Pertuzumab, Trastuzumab and Eribulin Dose Level 1 (D1: Pertuzumab: 840 mg/cycle 1 then 420 mg/cycle IV on day 1
  Trastuzumab: 8 mg/kg/cycle 1 then 6 mg/kg cycle IV on day 1
  Eribulin: 1.4 mg/m2/cycle IV on days 1 and 8 (D1)
  Cycle duration=21 days
  The Phase I run-in potentially evaluates 2 dose levels of eribulin in combination with pertuzumab and trastuzumab. Participants first receive antibody administration then eribulin. In the treatment phase, participants receive up to 6 cycles of combination therapy unless disease progression (PD) or withdrawal for other reasons (w/d). Participants who complete 6 cycles have the option to continue with antibody therapy only until PD or w/d in the extension phase.
Arm/Group | Phase I: Pertuzumab, Trastuzumab and Eribulin Dose Level 1 (D1
Number analyzed (Participants) | 6
mg/m^2 | 1.4

2. Primary Outcome: Dose Limiting Toxicity (DLT) [Phase I]
Description: A DLT was defined as an adverse event that (a) is deemed by the investigator to be probably or likely related with protocol therapy and (b) occurs during and/or begins during the first cycle of the study treatment, and (c) meets any of the following criteria: grade 4 hematologic toxicity with > 1 week of duration, grade 3 or 4 febrile neutropenia of any duration; or grade 3 or 4 non hematologic toxicity (excluding nausea, vomiting, and alopecia).
Time Frame: The observation period for DLTs was the 1st cycle of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: Pertuzumab, Trastuzumab and Eribulin Dose Level 1 (D1
Number analyzed (Participants) | 6
Participants | 0

3. Primary Outcome: Objective Response Rate (ORR) [Phase II]
Description: The objective response rate (ORR) was defined as the proportion of participants achieving complete response (CR) or partial response (PR) based on RECIST 1.1 criteria on treatment. Per RECIST 1.1 for target lesions: CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions.
Time Frame: Disease was evaluated radiologically at baseline and every 2 or 3 cycles in the treatment and extension phase, respectively. Median (range) treatment duration was 7(2-25) cycles for Cohort A and 4(3-18) cycles for Cohort B.
Population: The analysis dataset is comprised all enrolled Phase II patients.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Phase II Cohort A: Without Prior Pertuzumab Exposure | Phase II Cohort B: With Prior Pertuzumab Exposure
Number analyzed (Participants) | 19 | 7
proportion of participants | 0.26 [0.09 to 0.51] | 0.0 [0.0 to .41]

4. Secondary Outcome: Clinical Benefit Rate (CBR) [Phase II]
Description: The clinical benefit rate (CBR) was defined as the proportion of participants achieving complete response (CR), partial response (PR), or stable disease (SD) for 24 weeks or longer based on RECIST 1.1 criteria on treatment. Per RECIST 1.1 for target lesions: CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. PD is at least a 20% increase in sum LD of target lesions (smallest sum LD reference), new lesions, and/or unequivocal progression of existing non-target lesions. Stable disease (SD) is defined as any condition not meeting the above criteria.
Time Frame: as for outcome 3
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Phase II Cohort A: Without Prior Pertuzumab Exposure | Phase II Cohort B: With Prior Pertuzumab Exposure
Number analyzed (Participants) | 19 | 7
proportion of participants | .316 [.126 to .566] | .143 [.004 to .579]

5. Secondary Outcome: Progression-free Survival (PFS) [Phase II]
Description: Progression-free survival based on the Kaplan-Meier method is defined as the duration of time from study entry to documented disease progression (PD) or death. Per RECIST 1.1 criteria: progressive disease (PD) is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or equivocal progression of non-target lesions.(whichever occurs first).
Time Frame: Disease was evaluated radiologically at baseline, every 2 or 3 cycles in the treatment and extension phase, respectively, and every 9 weeks post-treatment until disease progression. Median follow-up in this study cohort was 15.6 months (up to 20).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II Cohort A: Without Prior Pertuzumab Exposure | Phase II Cohort B: With Prior Pertuzumab Exposure
Number analyzed (Participants) | 19 | 6
months | 6.9 [3.5 to 11] | 3 [2.1 to NA] — The upper confidence limit was not estimable based on the Kaplan-Meier method because of insufficient follow-up.

6. Secondary Outcome: Overall Survival (OS) [Phase II]
Description: Overall survival (OS) is defined as the time from the date of registration to the date of death, or censored at the date the participant was last known alive. OS is estimated based on the Kaplan-Meier method.
Time Frame: In long-term follow-up, participants were followed for survival every 6 months up to 1 year after treatment discontinuation. Median follow-up in this study cohort was 15.6 months (up to 20).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II Cohort A: Without Prior Pertuzumab Exposure | Phase II Cohort B: With Prior Pertuzumab Exposure
Number analyzed (Participants) | 19 | 6
months | 13.9 [11.2 to NA] — The upper confidence limit was not estimable based on the Kaplan-Meier method because of insufficient follow-up. | 7.4 [5.7 to NA] — The upper confidence limit was not estimable based on the Kaplan-Meier method because of insufficient follow-up.

7. Secondary Outcome: Grade 4 Treatment-Related Toxicity Rate
Description: Grade 4 treatment-related toxicity rate is the percentage of participants experiencing at least one treatment-related grade 4 adverse event (AE) of any type during the time of observation as reported on case report forms. 'Treatment-related' is a treatment attribution of possibly, probably or definite based on the NCI Common Toxicity Criteria for Adverse Events (CTCAE) version 4.
Time Frame: AEs were assessed every cycle on treatment. Median (range) treatment duration was 7(2-25) cycles for Cohort A and 4(3-18) cycles for Cohort B.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II Cohort A: Without Prior Pertuzumab Exposure | Phase II Cohort B: With Prior Pertuzumab Exposure
Number analyzed (Participants) | 19 | 7
percentage of participants | 10.5 [1.29 to 33.1] | 14.3 [0.4 to 57.9]

8. Post Hoc Outcome: 1-year Overall Survival
Description: 1-year overall survival is the probability of patients remaining alive 1 year from study entry estimated using Kaplan-Meier (KM) methods which censors patients at date of last follow-up.
Time Frame: as for outcome 6
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Phase II Cohort A: Without Prior Pertuzumab Exposure | Phase II Cohort B: With Prior Pertuzumab Exposure
Number analyzed (Participants) | 19 | 6
probability | 61.1 [42.3 to 88.3] | 50 [22.5 to 100]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were assessed each cycle throughout treatment from time of first dose and until outstanding adverse events are stable or resolved, if any. Median treatment duration (and thus average period for AE assessment) was 11.5 cycles, 7 cycles, 4 cycles for D1, Cohort A, Cohort B, respectively. Maximum treatment duration was 26 cycles, 25 cycles, 18 cycles for D1, Cohort A, Cohort B, respectively. Cycle length is 21 days/3 weeks.
Description: Maximum grade toxicity by type was first calculated. Serious AEs were defined as events with treatment-attribution of possible, probable or definite and grade 3 or higher per NCI Common Toxicity Criteria for Adverse Events (CTCAE) version 4. Other AEs included grade 3 or higher events unrelated to treatment and all grade 1-2 events.No further data is available to specify classification of other beyond the general term.
Arm/Group | Phase I: Dose Level 1 (D1) | Phase II Cohort A: Without Prior Pertuzumab Exposure | Phase II Cohort B: With Prior Pertuzumab Exposure
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/19 | 0/7
Serious Adverse Events (participants affected / at risk) | 4/6 | 7/19 | 4/7
Other Adverse Events (participants affected / at risk) | 6/6 | 18/19 | 5/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: Dose Level 1 (D1) (N=6) | Phase II Cohort A: Without Prior Pertuzumab Exposure (N=19) | Phase II Cohort B: With Prior Pertuzumab Exposure (N=7)
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 1 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 1 | 1
Neutrophil count decreased (Investigations) | 3 | 2 | 4
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: Dose Level 1 (D1) (N=6) | Phase II Cohort A: Without Prior Pertuzumab Exposure (N=19) | Phase II Cohort B: With Prior Pertuzumab Exposure (N=7)
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 1
Alanine aminotransferase increased (Investigations) | 0 | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 6 | 2
Anemia (Blood and lymphatic system disorders) | 0 | 2 | 2
Anorexia (Metabolism and nutrition disorders) | 1 | 3 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 3 | 1
Ataxia (Nervous system disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Bladder infection (Infections and infestations) | 0 | 0 | 1
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Bronchial infection (Infections and infestations) | 0 | 1 | 0
Cataract (Eye disorders) | 1 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 1 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Chills (General disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 7 | 3
Dizziness (Nervous system disorders) | 1 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Edema limbs (General disorders) | 0 | 1 | 0
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 1 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Facial nerve disorder (Nervous system disorders) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 11 | 0
Fatigue (General disorders) | 6 | 0 | 4
Fever (General disorders) | 0 | 0 | 2
Flu like symptoms (General disorders) | 0 | 1 | 0
Gait disturbance (General disorders) | 1 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Headache (Nervous system disorders) | 0 | 3 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 2 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Infusion related reaction (General disorders) | 1 | 1 | 0
Investigations - Other (Investigations) | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 2 | 0
Memory impairment (Nervous system disorders) | 1 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 2 | 3 | 0
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 8 | 2
Neutrophil count decreased (Investigations) | 2 | 3 | 0
Pain (General disorders) | 2 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Palpitations (Cardiac disorders) | 0 | 1 | 0
Paronychia (Infections and infestations) | 1 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 6 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 6 | 2
Platelet count decreased (Investigations) | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Rash pustular (Infections and infestations) | 0 | 2 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Upper respiratory infection (Infections and infestations) | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 1 | 1
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 4 | 0
Watering eyes (Eye disorders) | 0 | 0 | 1
Weight loss (Investigations) | 1 | 0 | 0
White blood cell decreased (Investigations) | 0 | 3 | 0

LIMITATIONS AND CAVEATS:
The study is limited as it was terminated early due to slow accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No